CLINICAL TRIAL: NCT02326116
Title: Investigating the Role of Tracheal Traction Exercises (TTE) in Reducing Dysphagia Following Anterior Cervical Surgery
Brief Title: TTE and Dysphagia in Anterior Cervical Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 54543
Record Dates: First submitted 2014-12-20; First posted 2014-12-25 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Trachael Traction Exercises
  Interventions: Other: Trachael Preparation Education
- Group 2 (Placebo Comparator): Trachael Massage
  Interventions: Other: Trachael Preparation Education

INTERVENTIONS:
Other: Trachael Preparation Education

SUMMARY:
The purpose of this study is to evaluate if Tracheal Traction Exercises (TTE) performed prior to anterior cervical spine surgery can result in a decreased rate of dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* Elective Anterior cervical spine surgery (C2-C7) for degenerative disc disease or myelopathy

Exclusion Criteria:

* More than four levels of fusion
* Trauma or urgent cases of anterior cervical spine surgery
* Prior anterior cervical spine surgery (a known risk factor for dysphagia),
* Prior neck surgery (eg. Thyroidectomy)
* Tumors
* Infections
* Neurological disorders that can predispose to dysphagia such as Parkinson's, Cerebrovascular Accidents (CVA), Alzheimer's and Amyotrophic Lateral Sclerosis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-11; Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
SWAL-QOL | 12 months
  30% difference in dysphagia as quantified by the SWAL-QOL (validated measure of dysphagia)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States